CLINICAL TRIAL: NCT01609387
Title: Postoperative Vitamin Supplementation in Morbidly Obese Patient
Brief Title: Postoperative Vitamin Supplementation in Morbidly Obese Patient (VITAAL Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Jens Homan, Investigator, Rijnstate Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LTC 745
Record Dates: First submitted 2011-09-15; First posted 2012-06-01 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Obesity; Vitamin Deficiency
Keywords: Vitamine; mineral; obese patients; Vitamine en mineral shortage in obese patients
MeSH Terms: conditions — Obesity; Avitaminosis; Calcinosis | interventions — Tocopherols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Gastric Banding new vitamins (Experimental): Randomization between optimal multivitamins for bariatric surgery and normal over the counter multivitamins (in Gastric Band patients)
  Interventions: Dietary Supplement: Fit For me
- Gastric Banding current vitamins (Active Comparator): Randomization between optimal multivitamins for bariatric surgery and normal over the counter multivitamins (in Gastric Band patients)
  Interventions: Dietary Supplement: Davitamon
- RYGB new vitamins (Experimental): Randomization between optimal multivitamins for bariatric surgery and normal over the counter multivitamins (in RYGB patients
  Interventions: Dietary Supplement: Fit For me
- RYGB current vitamins (Active Comparator): Randomization between optimal multivitamins for bariatric surgery and normal over the counter multivitamins (in RYGB patients)
  Interventions: Dietary Supplement: Davitamon
- Gastric sleeve new vitamins (Experimental): Randomization between optimal multivitamins for bariatric surgery and normal over the counter multivitamins (in Gastric Sleeve patients)
  Interventions: Dietary Supplement: Fit For me
- Gastric sleeve current vitamins (Active Comparator): Randomization between optimal multivitamins for bariatric surgery and normal over the counter multivitamins (in Gastric Sleeve patients)
  Interventions: Dietary Supplement: Davitamon

INTERVENTIONS:
Dietary Supplement: Fit For me
  Arms: Gastric Banding new vitamins; Gastric sleeve new vitamins; RYGB new vitamins
Dietary Supplement: Davitamon
  Arms: Gastric Banding current vitamins; Gastric sleeve current vitamins; RYGB current vitamins

SUMMARY:
This study is a double blind randomized controlled trial.

DETAILED DESCRIPTION:
Based on evidence-based literature on vitamins and minerals, there is a cooperation of a manufacturer multivitamin specifically designed for patients with a gastric band and Roux-en-Y gastric bypass (RYGB). These preparations are the proportions adjusted so that the risk of shortages should decrease and on the other hand, excessive levels of nutrients should be avoided. Main objective of this study is to examine whether these new supplements in particular the number of deficiencies in iron, vitamin B12 and vitamin D can be reduced.

ELIGIBILITY:
Inclusion Criteria:

* Patients on the waiting list for RYGB or gastric band and meets
* Age between 18-65 years

Exclusion Criteria:

1. Creatinine > 150micromol / L
2. Liver enzymes > 2 times the upper limit
3. Previous surgery on the gastrointestinal tract
4. Intercurrerence disease
5. Gastrointestinal Diseases
6. Psychiatric illness
7. Drugs that affect bone metabolism
8. Known pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-07; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Reduction of iron deficiency in obese patients | one year

SECONDARY OUTCOMES:
Reduction of vitamin D and vitamin B12 deficiency | one year

CONTACTS AND LOCATIONS:
Overall Officials: Frits Berends, MD,PhD, Principal Investigator — Rijnstate Arnhem
Locations (1):
- Rijnstate Hospital, Arnhem, Wagnerlaan 55, Netherlands

REFERENCES:
- [Derived] Heusschen L, Schijns W, Ploeger N, Deden LN, Hazebroek EJ, Berends FJ, Aarts EO. The True Story on Deficiencies After Sleeve Gastrectomy: Results of a Double-Blind RCT. Obes Surg. 2020 Apr;30(4):1280-1290. doi: 10.1007/s11695-019-04252-1. PMID 31776782